CLINICAL TRIAL: NCT00585481
Title: Incidence of Severe Respiratory Syncytial Virus Infections in Preterm Brazilian Children - BREVI (Brazilian Respiratory Virus in Premature Infants) Study
Brief Title: Incidence of Severe Respiratory Syncytial Virus Infections in Preterm Brazilian Children
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Statistika Consultoria Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: A07-006
Record Dates: First submitted 2007-12-22; First posted 2008-01-03 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Respiratory Syncytial Viruses; Respiratory Tract Infection
Keywords: Epidemiological Study; Incidence of severe Respiratory Syncytial Virus; Preterm Brazilian children
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white cells and nasopharyngal aspirate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All subjects will perform samples collection for RSV analysis. Subject's enrolled in Porto Alegre's site will perform lung function tests.
  Interventions: Procedure: Samples collection for viral diagnosis; Procedure: Lung Function Analysis

INTERVENTIONS:
Procedure: Samples collection for viral diagnosis — At Enrollment and Termination Visits all subjects will have phlebotomy performed for RSV antibody levels (3 mL of blood).
  Subjects diagnosed with an LRTI during the study will have a nasopharyngeal lavage (NPL) for viral diagnosis. Phlebotomy for antibody levels will be performed if the current episode represents the first LRTI since study enrollment.
Procedure: Lung Function Analysis — Subjects enrolled in one study site (located in Porto Alegre city) will perform Lung Function Analysis. First measurement will be performed up to Visit 6 and repeated at Termination Visit. Measurements collected in the first analysis will include respiratory compliance and resistance by passive deflation pressure - volume curve, lung volumes by gas dilution method (washout with SF6), lung clearance index with SF6, and maximal flows (rapid thoracic compression from raised volumes).

SUMMARY:
The primary objective of this study is to determine the incidence of severe RSV LRTI requiring hospitalization among infants born < 35 weeks gestational age for one year of follow-up.

DETAILED DESCRIPTION:
This is an epidemiologic study of the incidence of severe RSV LRTI among Brazilian children born <35WGA. The study will enroll competitively 350 subjects from 3 sites in Brazil. Preterm children will be identified after birth and up to 72 hours after hospital discharge and followed for one year after the enrollment. Subjects will be seen monthly for the first 6 months and bimonthly until one year of follow-up. At each visit, a medical and social history will be updated and a physical examination will be performed. Legal representative will notify study personnel in the event of a respiratory illness or hospital admission at which time the subject will be seen by an investigator. Children with LRTI diagnosed by physical examination will have viral diagnostic tests performed. Subjects with a LRTI not requiring hospitalization will be followed by telephone weekly until illness resolution. Hospitalized children with a LRTI will be followed daily while hospitalized and followed by telephone until illness resolution. All medical interventions and outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male and female infants that were born <35 weeks gestational age
* The inclusion must be done during the following period:

  * 24 hours prior confirmed maternity hospital discharge date, or
  * Up to 72 hours after documented maternity hospital discharge date. In this case, RSV rapid test must be performed and subjects should be enrolled only if the results is negative.
* Less than 6 months of age at screening
* Born into or transferred to a participating hospital
* Able to receive follow-up medical care at the participating site and provide information during the follow-up period
* The legal representative is capable of understanding and complying with parameters as outlined in the protocol and able and willing to participate in this study, by signing the informed consent approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), after all the aspects of the study that might be relevant for his/her decision to participate are explained and all his/her questions and doubts are elucidated, and prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* RSV infection prior inclusion.
* Receipt of palivizumab or other immunoglobulin preparation containing RSV specific antibodies (i.e. RSV hyperimmunoglobulin, polyclonal intravenous immunoglobulin, cytomegalovirus hyperimmunoglobulin, varicella-zoster hyperimmunoglobulin)

Max Age: 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants < 35 wGA born into or transferred to a participating hospital meeting all of the inclusion criteria and none of the exclusion criteria specified in the protocol will be selected to participate. Subjects will be identified in the NICU or newborn nursery and enrolled in the study 24 hours prior to confirmed hospital discharge or up to 72 hours after maternity hospital discharge date.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of severe RSV LRTI requiring hospitalization among infants born <35 weeks gestational age for one year. | 1 Year

SECONDARY OUTCOMES:
To evaluate the risk and protective factors for severe RSV LRTI in preterm Brazilian infants. | 1 Year
To describe the seasonality of RSV infection in three cities in Brazil. | 1 Year
To compare the incidence of wheezing episodes by 12 months after maternity hospital discharge among children with and without RSV LRTI. | 1 Year
To evaluate the difference in lung function among children with and without RSV LRTI within the first year after maternity hospital discharge. Only children enrolled at one participating site will be evaluated with lung function analysis. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Lino Rodrigues, MD, Study Chair — Abbott Laboratórios do Brasil Ltda.
Locations (2):
- Brazil (2):
  - Site Ref # / Investigator 6185, Curitiba, Paraná
  - Site Ref # / Investigator 6189, Ribeirão Preto, São Paulo

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=23151&CFID